CLINICAL TRIAL: NCT06418815
Title: Effect of Concept Map on Nursing Students' Ability to Assess Toxic Stress in Newborns: A Randomized Controlled Trial
Brief Title: Concept Map on Toxic Stress in Newborns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Aylin PEKYİGİT, Research Assistant PhD, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CKU12
Record Dates: First submitted 2024-04-24; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Nursing Education; Newborn
Keywords: Concept map; Nursing education; Toxic stress; Newborn

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concept Map Group (Experimental): The intervention group will create a concept map regarding neonatal toxic stress.
  Interventions: Other: Concept map group
- Control Group (No Intervention): During the application process of the research, knowledge tests will be applied as pre-test and post-test

INTERVENTIONS:
Other: Concept map group — The intervention group will create a concept map regarding neonatal toxic stress.
  Arms: Concept Map Group

SUMMARY:
This study will be conducted as a single-blind randomized control group intervention trial to examine the effect of using concept maps on the students' knowledge levels about toxic stress in newborns, which is explained to second-year nursing students.

DETAILED DESCRIPTION:
The Newborn Toxic Stress Knowledge Test (1st Test) will be administered to intervention and control group students who agree to participate in the research, before the 4-hour High Risk Newborn theoretical lecture. Training on Toxic Stress in Newborns will be given to both groups, and then a post-training knowledge test (2nd Test) will be administered. The initiative group will be composed of students who apply concept maps and make in-class maintenance plans after theoretical training. The control group will consist of students who receive theoretical training and implement in-class care plans. After the concept map application, a knowledge test will be applied again (3rd Test).

The data of the research will be collected with the Personal Information Form and Newborn Toxic Stress Information Test.

The personal information form was prepared by the researchers. In shape; There are questions about the student's age, gender, secondary school graduation status, whether they choose the nursing profession willingly, whether they consider the nursing profession suitable for themselves, whether they have heard the term concept map and whether they have applied concept map.

Newborn Toxic Stress Information Test was prepared by researchers. The test consists of 25 multiple choice questions. It consists of true, false and I don't know options.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the course
* Had not taken this course before
* Accepted to participate in the research

Exclusion Criteria:

* Have any records of absence
* Taken this course before
* Graduate of health vocational high school

Ages: 19 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2024-05-13 (Estimated); Study Completion 2024-06-06 (Estimated)

PRIMARY OUTCOMES:
Differences of knowledge scores between groups | The first knowledge test (pre-test) will be given before class in the first week. Two knowledge tests will be administered for the final test. Total duration is 4 weeks.
  First, second and thirth knowledge tests will be applied to measure the level of knowledge. The student can get a minimum of 0 and a maximum of 100 from the knowledge test. Higher scores mean better results.

REFERENCES:
- [Background] Sand-Jecklin K. The impact of active/cooperative instruction on beginning nursing student learning strategy preference. Nurse Educ Today. 2007 Jul;27(5):474-80. doi: 10.1016/j.nedt.2006.08.006. Epub 2006 Oct 9. PMID 17030077
- [Background] Gul RB, Boman JA. Concept mapping: A strategy for teaching and evaluation in nursing education. Nurse Educ Pract. 2006 Jul;6(4):199-206. doi: 10.1016/j.nepr.2006.01.001. Epub 2006 Feb 28. PMID 19040878
- [Background] Baliga SS, Walvekar PR, Mahantshetti GJ. Concept map as a teaching and learning tool for medical students. J Educ Health Promot. 2021 Jan 28;10:35. doi: 10.4103/jehp.jehp_146_20. eCollection 2021. PMID 33688544